CLINICAL TRIAL: NCT01872975
Title: A Randomized Phase III Clinical Trial Evaluating Post-Mastectomy Chestwall and Regional Nodal XRT and Post-Lumpectomy Regional Nodal XRT in Patients With Positive Axillary Nodes Before Neoadjuvant Chemotherapy Who Convert to Pathologically Negative Axillary Nodes After Neoadjuvant Chemotherapy
Brief Title: Standard or Comprehensive Radiation Therapy in Treating Patients With Early-Stage Breast Cancer Previously Treated With Chemotherapy and Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NSABP Foundation Inc (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Radiation Therapy Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSABP-B-51; NCI-2012-03198 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); U10CA012027 (NIH)
Record Dates: First submitted 2013-06-03; First posted 2013-06-07 (Estimated); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Stage IB Breast Cancer; Stage II Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1A Lumpectomy: no regional nodal XRT with WBI (Active Comparator): Lumpectomy patients undergo whole breast radiation therapy using IMRT or 3D-CRT once daily 5 days a week for 5 weeks followed by a radiation therapy boost to the lumpectomy cavity once daily 5 days a week for 1-1/2 weeks.
  Interventions: Radiation: WBI
- Group 1B Mastectomy: No regional nodal or chestwall XRT (No Intervention): Mastectomy patients do not undergo radiation therapy.
- Group 2A lumpectomy: Regional nodal XRT with WBI (Experimental): Lumpectomy patients undergo regional nodal radiation therapy with whole breast radiation therapy using IMRT or 3D-CRT once daily 5 days a week for 5 weeks followed by a radiation therapy boost to the lumpectomy cavity once daily 5 days a week for 1-1/2 weeks.
  Interventions: Radiation: regional nodal XRT; Radiation: WBI
- Group 2B Mastectomy: Regional nodal XRT and chestwall XRT (Experimental): Mastectomy patients undergo regional nodal radiation therapy using IMRT or 3D-CRT once daily 5 days a week for 5 weeks.
  Interventions: Radiation: regional nodal XRT; Radiation: chestwall XRT

INTERVENTIONS:
Radiation: regional nodal XRT
  Other Names: XRT: External radiotherapy
  Arms: Group 2A lumpectomy: Regional nodal XRT with WBI; Group 2B Mastectomy: Regional nodal XRT and chestwall XRT
Radiation: chestwall XRT
  Other Names: XRT: External radiotherapy
  Arms: Group 2B Mastectomy: Regional nodal XRT and chestwall XRT
Radiation: WBI
  Other Names: Whole Breast Irradiation (WBI)
  Arms: Group 1A Lumpectomy: no regional nodal XRT with WBI; Group 2A lumpectomy: Regional nodal XRT with WBI

SUMMARY:
This randomized phase III trial studies standard or comprehensive radiation therapy in treating patients with early-stage breast cancer who have undergone surgery. Radiation therapy uses high-energy x rays to kill tumor cells. It is not yet known whether comprehensive radiation therapy is more effective than standard radiation therapy in treating patients with breast cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

To evaluate whether the addition of chest wall + regional nodal radiation therapy (XRT) after mastectomy or breast + regional nodal XRT after breast conserving surgery will significantly reduce the rate of events for invasive breast cancer recurrence-free interval (IBC-RFI) in patients who present with histologically positive axillary nodes but convert to histologically negative axillary nodes following neoadjuvant chemotherapy.

SECONDARY OBJECTIVES:

I. To evaluate whether the addition of chest wall + regional nodal XRT after mastectomy or breast + regional nodal XRT after breast conserving surgery will significantly prolong overall survival (OS) in patients who present with histologically positive axillary nodes but convert to histologically negative axillary nodes following neoadjuvant chemotherapy.

II. To evaluate whether the addition of chest wall + regional nodal XRT after mastectomy or breast + regional nodal XRT after breast conserving surgery will significantly reduce the rates of events for local-regional recurrence-free interval (LRRFI) in patients who present with histologically positive axillary nodes but convert to histologically negative axillary nodes following neoadjuvant chemotherapy.

III. To evaluate whether the addition of chest wall + regional nodal XRT after mastectomy or breast + regional nodal XRT after breast conserving surgery will significantly reduce the rate of events for distant recurrence-free interval (DRFI) in patients who present with histologically positive axillary nodes but convert to histologically negative axillary nodes following neoadjuvant chemotherapy.

IV. To compare the rates of disease-free survival (DFS)-ductal carcinoma in situ (DCIS) by treatment arm.

V. To compare the rates of second primary cancer (SPC) by treatment arm.

VI. To compare the effect of adding XRT on the cosmetic outcomes in mastectomy patients who have had reconstruction.

VII. To compare the effect of adding XRT on quality of life including arm problems, lymphedema, pain, and fatigue.

VIII. To evaluate the toxicity associated with each of the radiation therapy regimens.

IX. To determine whether computed tomography (CT)-based conformal methods (intensity-modulated radiation therapy [IMRT] and 3-dimensional conformal radiation therapy [3DCRT]) for chestwall + regional nodal XRT post mastectomy and regional nodal XRT with breast XRT following breast conserving surgery are feasible in a multi-institutional setting and whether dose-volume analyses can be established to assess treatment adequacy and to develop normal tissue complication probabilities (NTCP) for the likelihood of toxicity.

X. To compare the effect of XRT in patients receiving mastectomy and in patients receiving lumpectomy.

XI. To examine the role of proliferation measures as a prognosticator for patients with residual disease after neoadjuvant chemotherapy.

XII. To develop predictors of the degree of reduction in local regional recurrence (LRR).

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM 1: Patients are assigned to 1 of 2 treatment groups.

GROUP 1A: Lumpectomy patients undergo whole breast radiation therapy using IMRT or 3DCRT once daily 5 days a week for 5 weeks followed by a radiation therapy boost to the lumpectomy cavity once daily 5 days a week for 1-1/2 weeks.

GROUP 1B: Mastectomy patients do not undergo radiation therapy.

ARM 2: Patients are assigned to 1 of 2 treatment groups.

GROUP 2A: Lumpectomy patients undergo regional nodal radiation therapy with whole breast radiation therapy using IMRT or 3DCRT once daily 5 days a week for 5 weeks followed by a radiation therapy boost to the lumpectomy cavity once daily 5 days a week for 1-1/2 weeks.

GROUP 2B: Mastectomy patients undergo regional nodal radiation therapy and chestwall XRT using IMRT or 3DCRT once daily 5 days a week for 5 weeks.

All patients also receive systemic therapy as planned (hormonal therapy for patients with hormone-receptor positive breast cancer and trastuzumab or other anti-human epidermal growth factor receptor 2 [HER2] therapy for patients with breast cancer that is HER2-positive).

After completion of study treatment, patients are followed up at 6, 12, 18, and 24 months and then yearly for 8 years.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have signed and dated an Institutional Review Board (IRB)-approved consent form that conforms to federal and institutional guidelines
* The patient must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Patient must have clinically T1-3, N1 breast cancer at the time of diagnosis (before neoadjuvant therapy); clinical axillary nodal involvement can be assessed by palpation, ultrasound, CT scan, magnetic resonance imaging (MRI), positron emission tomography (PET) scan, or PET/CT scan
* Patient must have had pathologic confirmation of axillary nodal involvement at presentation (before neoadjuvant therapy) based on either a positive fine needle aspirate (FNA) (demonstrating malignant cells) or positive core needle biopsy (demonstrating invasive adenocarcinoma); the FNA or core needle biopsy can be performed either by palpation or by image guidance; documentation of axillary nodal positivity by sentinel node biopsy (before neoadjuvant therapy) is not permitted
* Patients must have had estrogen receptor (ER) analysis performed on the primary breast tumor before neoadjuvant therapy according to current American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guideline recommendations for hormone receptor testing; if negative for ER, assessment of progesterone receptor (PgR) must also be performed according to current ASCO/CAP guideline recommendations for hormone receptor testing (http://www.asco.org)
* Patients must have had HER2 testing performed on the primary breast tumor before neoadjuvant chemotherapy according to the current ASCO/CAP guideline recommendations for human epidermal growth factor receptor 2 testing in Breast Cancer (http://www.asco.org); patients who have a primary tumor that is either HER2-positive or HER2-negative are eligible
* Patient must have completed a minimum of 8 weeks of standard neoadjuvant chemotherapy consisting of an anthracycline and/or taxane-based regimen
* For patients who receive adjuvant chemotherapy after surgery, a maximum of 12 weeks of intended chemotherapy may be administered but must be completed before randomization; (if treatment delays occur, chemotherapy must be completed within 14 weeks); the dose and schedule of the adjuvant chemotherapy are at the investigator's discretion; Note: It is preferred that all intended chemotherapy be administered in the neoadjuvant setting
* Patients with HER2-positive tumors must have received neoadjuvant anti-HER2 therapy (either with all or with a portion of the neoadjuvant chemotherapy regimen), unless medically contraindicated
* At the time of definitive surgery, all removed axillary nodes must be histologically free from cancer; acceptable procedures for assessment of axillary nodal status at the time of surgery include:

  * Axillary node dissection
  * Sentinel node biopsy alone or
  * Sentinel node biopsy followed by axillary node dissection
  * Note: Patients are eligible whether there is residual invasive carcinoma in the surgical breast specimen or whether there is evidence of pathologic complete response; patients who are found to be pathologically node-positive at the time of surgery, based on sentinel node biopsy alone, are candidates for A011202, a study developed by the Alliance in Oncology, an NCI Cooperative Group; if A011202 is open at the investigator's institution, patients should be approached about participating in the A011202 study
* Patients with pathologic staging of ypN0(i+) or ypN0(mol+) are eligible (Note: Postneoadjuvant therapy is designated with a "yp" prefix.)
* Patient who have undergone either a total mastectomy or a lumpectomy are eligible
* For patients who undergo lumpectomy, the margins of the resected specimen or re-excision must be histologically free of invasive tumor and DCIS as determined by the local pathologist; additional operative procedures may be performed to obtain clear margins; if tumor is still present at the resected margin after re-excision(s), the patient must undergo total mastectomy to be eligible; (patients with margins positive for lobular carcinoma in situ [LCIS] are eligible without additional resection)
* For patients who undergo mastectomy, the margins must be histologically free of residual (microscopic or gross) tumor
* The interval between the last surgery for breast cancer (including re-excision of margins) and randomization must be no more than 70 days; also, if adjuvant chemotherapy was administered, the interval between the last chemotherapy treatment and randomization must be no more than 70 days
* The patient must have recovered from surgery with the incision completely healed and no signs of infection
* If adjuvant chemotherapy was administered, chemotherapy-related toxicity that may interfere with delivery of radiation therapy should have resolved

Exclusion Criteria:

* Definitive clinical or radiologic evidence of metastatic disease
* T4 tumors including inflammatory breast cancer
* Documentation of axillary nodal positivity before neoadjuvant therapy by sentinel node biopsy alone
* N2 or N3 disease detected clinically or by imaging
* Patients with histologically positive axillary nodes post neoadjuvant therapy
* Patients with microscopic positive margins after definitive surgery
* Synchronous or previous contralateral invasive breast cancer or DCIS; (patients with synchronous and/or previous contralateral LCIS are eligible)
* Any prior history, not including the index cancer, of ipsilateral invasive breast cancer or ipsilateral DCIS treated with radiation therapy; (patients with synchronous or previous ipsilateral LCIS are eligible)
* History of non-breast malignancies (except for in situ cancers treated only by local excision and basal cell and squamous cell carcinomas of the skin) within 5 years prior to randomization
* Any radiation therapy for the currently diagnosed breast cancer prior to randomization
* Any continued use of sex hormonal therapy, e.g., birth control pills, ovarian hormone replacement therapy; patients are eligible if these medications are discontinued prior to randomization
* Prior breast or thoracic radiation therapy (RT) for any condition
* Active collagen vascular disease, specifically dermatomyositis with a creatinine phosphokinase (CPK) level above normal or with an active skin rash, systemic lupus erythematosus, or scleroderma
* Pregnancy or lactation at the time of study entry; (Note: Pregnancy testing must be performed within 2 weeks prior to randomization according to institutional standards for women of childbearing potential)
* Other non-malignant systemic disease that would preclude the patient from receiving study treatment or would prevent required follow-up
* Psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude the patient from meeting the study requirements

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1636 (Estimated)
Dates: Start 2013-08; Primary Completion 2023-09-14 (Actual); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
IBC-RFI | Time from randomization until invasive local, regional, or distant recurrence, or death from breast cancer, assessed up to 10 years

SECONDARY OUTCOMES:
OS | Time from randomization to death from any cause, assessed up to 10 years
LRRFI | Time from randomization to recurrence of primary cancer w/in breast or lymph nodes in ipsilateral axilla, infraclavicular fossa, or ipsilateral internal mammary chain w/out evidence distant disease, or death due to breast cancer, assessed up to 10 years
DRFI | Time from randomization to the development of tumor in all areas beyond local or regional limits, or death due to breast cancer, assessed up to 10 years
DFS-DCIS | Time from randomization to local recurrence post-mastectomy/in ipsilateral breast post-lumpectomy, regional/distant recurrence, contralateral disease, second primary cancer, or death from any cause prior to recurrence or SPC, assessed up to 10 years
Time to SPC | Time from randomization to the development of a second primary invasive cancer of any site excluding squamous and basal cell carcinoma of the skin, assessed up to 10 years
Effect of radiation therapy on cosmetic outcome in mastectomy and lumpectomy patients as assessed by quality of life questionnaire | Assessed prior to randomization, 3 months or at end of RT, and 6, 12, and 24 months from randomization
Frequencies of adverse events graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Up to 30 days after completion of study treatment
Molecular predictors of recurrence | Tissue samples collected within 90 days after randomization
  To test the prognostic role of gene expression profiles in residual tumor tissue and to develop predictors of the degree of reduction of loco-regional recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (514):
- United States (489):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Arizona Breast Cancer Specialists-Gilbert, Gilbert, Arizona
  - Arizona Center for Cancer Care-Peoria, Peoria, Arizona
  - Arizona Breast Cancer Specialists-Phoenix, Phoenix, Arizona
  - Arizona Breast Cancer Specialists-Scottsdale, Scottsdale, Arizona
  - Arizona Center for Cancer Care-Surprise, Surprise, Arizona
  - Arizona Oncology Associates-West Orange Grove, Tucson, Arizona
  - The University of Arizona Medical Center-University Campus, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Mills - Peninsula Hospitals, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Eden Hospital Medical Center, Castro Valley, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Epic Care-Dublin, Dublin, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - California Cancer Center - North Fresno, Fresno, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - City of Hope Antelope Valley, Lancaster, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Hoag Memorial Hospital, Newport Beach, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Saint Joseph Hospital - Orange, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Desert Regional Medical Center, Palm Springs, California
  - Huntington Memorial Hospital, Pasadena, California
  - Pomona Valley Hospital Medical Center, Pomona, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Sutter General Hospital, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Naval Medical Center -San Diego, San Diego, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - City of Hope South Pasadena, South Pasadena, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Saint Helena Hospital, St. Helena, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Memorial Hospital Colorado Springs, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - The Shaw Regional Cancer Center, Edwards, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Middlesex Hospital, Middletown, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Florida Hospital Cancer Institute Altamonte, Altamonte Springs, Florida
  - John Fitzgerald Kennedy Medical Center, Atlantis, Florida
  - Morton Plant Hospital, Clearwater, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - University of Florida, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Jackson Memorial Hospital-Holtz Children's Hospital, Miami, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - South Miami Hospital, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - 21st Century Oncology-Palatka, Palatka, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - Tanner Medical Center/Carrollton, Carrollton, Georgia
  - Dekalb Medical Center, Decatur, Georgia
  - Memorial University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Queen's Medical Center, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Leeward, ‘Ewa Beach, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - AMITA Health Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Edward Hospital/Cancer Center?Plainfield, Plainfield, Illinois
  - SwedishAmerican Regional Cancer Center/ACT, Rockford, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Saint Vincent Anderson Regional Hospital/Cancer Center, Anderson, Indiana
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - Community Cancer Center East, Indianapolis, Indiana
  - Community Cancer Center South, Indianapolis, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Community Cancer Center North, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Saint Elizabeth Medical Center South, Edgewood, Kentucky
  - Saint Elizabeth Fort Thomas, Fort Thomas, Kentucky
  - Norton Hospital Pavilion and Medical Campus, Louisville, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Norton Suburban Hospital and Medical Campus, Louisville, Kentucky
  - Owensboro Health Mitchell Memorial Cancer Center, Owensboro, Kentucky
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Woman's Hospital, Baton Rouge, Louisiana
  - Mary Bird Cancer Center/Saint Tammany Parish, Covington, Louisiana
  - Mary Bird Perkins Cancer Center/Terrebonne General Medical Center, Houma, Louisiana
  - Ochsner Medical Center Kenner, Kenner, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Medical Center- Scarborough Campus, Scarborough, Maine
  - Anne Arundel Medical Center, Annapolis, Maryland
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Upper Chesapeake Medical Center, Bel Air, Maryland
  - Central Maryland Radiation Oncology in Howard County, Columbia, Maryland
  - Tate Cancer Center, Glen Burnie, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Saint Anne's Hospital, Fall River, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Henry Ford Cancer Institute¿Downriver, Brownstown, Michigan
  - 21st Century Oncology-Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Beaumont Hospital-Dearborn, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - McLaren Cancer Institute-Central Michigan, Mount Pleasant, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Assarian Cancer Center, Novi, Michigan
  - McLaren Cancer Institute-Owosso, Owosso, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Providence Hospital-Southfield Cancer Center, Southfield, Michigan
  - 21st Century Oncology-Troy, Troy, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Mayo Clinic Health System in Albert Lea, Albert Lea, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Mayo Clinic Radiation Therapy-Northfield, Northfield, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Baptist Memorial Hospital-Desoto, Southhaven, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Siteman Cancer Center - Saint Peters, City of Saint Peters, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Barnes-Jewish West County Hospital, Creve Coeur, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - The University of Kansas Cancer Center-North, Kansas City, Missouri
  - The University of Kansas Cancer Center-Lee's Summit, Lee's Summit, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Saint Anthony's Medical Center, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Concord Hospital, Concord, New Hampshire
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Elliot Hospital, Manchester, New Hampshire
  - Memorial Sloan Kettering Cancer Center at Basking Ridge, Basking Ridge, New Jersey
  - Ocean Medical Center, Brick, New Jersey
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - The Valley Hospital-Luckow Pavilion, Paramus, New Jersey
  - Capital Health Medical Center-Hopewell, Pennington, New Jersey
  - Riverview Medical Center/Booker Cancer Center, Red Bank, New Jersey
  - Valley Hospital, Ridgewood, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Sparta Cancer Treatment Center, Sparta, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Valley Health System-Hematology/Oncology, Westwood, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Lovelace Radiation Oncology, Albuquerque, New Mexico
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - Memorial Medical Center - Las Cruces, Las Cruces, New Mexico
  - Christus Saint Vincent Regional Cancer Center, Santa Fe, New Mexico
  - New York-Presbyterian/Brooklyn Methodist Hospital, Brooklyn, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Putnam Hospital Center, Carmel, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Vassar Brothers Fishkill Radiation Oncology Center, Fishkill, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Ulster Radiation Oncology Center, Kingston, New York
  - Columbia University/Herbert Irving Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Vassar Brothers Medical Center, Poughkeepsie, New York
  - Rochester General Hospital, Rochester, New York
  - Pluta Cancer Center, Rochester, New York
  - Memorial Sloan Kettering Rockville Centre, Rockville Centre, New York
  - Memorial Sloan Kettering Sleepy Hollow, Sleepy Hollow, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute-Pineville, Charlotte, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute-University, Charlotte, North Carolina
  - Carolinas HealthCare System NorthEast, Concord, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - CaroMont Regional Medical Center, Gastonia, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Matthews Radiation Oncology Center, Matthews, North Carolina
  - Carolinas HealthCare System Union, Monroe, North Carolina
  - South Atlantic Radiation Oncology, Supply, North Carolina
  - Coastal Carolina Radiation Oncology, Wilmington, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Akron General Medical Center, Akron, Ohio
  - Summa Barberton Hospital, Barberton, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Geaugra Hospital, Chardon, Ohio
  - University of Cincinnati/Barrett Cancer Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Summa Health Center at Lake Medina, Medina, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - Southwest General Health Center Ireland Cancer Center, Middleburg Heights, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - University Pointe, West Chester, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Willamette Valley Cancer Center, Eugene, Oregon
  - Compass Oncology Rose Quarter, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Mid-Columbia Medical Center/Celilo Cancer Center, The Dalles, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Northeast Radiation Oncology Center, Dunmore, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - The Regional Cancer Center, Erie, Pennsylvania
  - Fox Chase Cancer Center Buckingham, Furlong, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - PinnacleHealth Cancer Center-Community Campus, Harrisburg, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Holy Redeemer Hospital and Medical Center, Meadowbrook, Pennsylvania
  - Intercommunity Cancer Center, Monroeville, Pennsylvania
  - UPMC-Coraopolis/Heritage Valley Radiation Oncology, Moon Township, Pennsylvania
  - Allegheny Valley Hospital, Natrona Heights, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Wexford Health and Wellness Pavilion, Wexford, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Radiation Oncology Associates Incorporated, Providence, Rhode Island
  - Women and Infants Hospital, Providence, Rhode Island
  - Kent County Hospital, Warwick, Rhode Island
  - Roper Hospital, Charleston, South Carolina
  - Bon Secours Saint Francis Hospital, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Georgetown Hospital System, Georgetown, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - The Radiation Oncology Center-Hilton Head/Bluffton, Hilton Head Island, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Lexington Medical Center, West Columbia, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - The West Clinic - Wolf River, Germantown, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Texas Cancer Center, Abilene, Texas
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Texas Oncology-Arlington South, Arlington, Texas
  - Texas Oncology-Austin Midtown, Austin, Texas
  - Texas Oncology - Central Austin Cancer Center, Austin, Texas
  - Texas Oncology - South Austin Cancer Center, Austin, Texas
  - Texas Oncology Bedford, Bedford, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Texas Oncology-Flower Mound, Flower Mound, Texas
  - The Klabzuba Cancer Center, Fort Worth, Texas
  - Memorial Hermann Memorial City Medical Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - The Methodist Hospital System, Houston, Texas
  - MD Anderson Regional Care Center-Katy, Houston, Texas
  - Doctor's Hospital of Laredo, Laredo, Texas
  - Covenant Medical Center-Lakeside, Lubbock, Texas
  - University Medical Center, Lubbock, Texas
  - Texas Tech University Health Sciences Center-Lubbock, Lubbock, Texas
  - MD Anderson Regional Care Center-Bay Area, Nassau Bay, Texas
  - Texas Oncology-Plano West, Plano, Texas
  - Scott and White Healthcare Round Rock, Round Rock, Texas
  - Texas Oncology - Round Rock Cancer Center, Round Rock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Texas Cancer Center-Sherman, Sherman, Texas
  - MD Anderson Regional Care Center-Sugar Land, Sugar Land, Texas
  - Texas Oncology Cancer Center Sugar Land, Sugar Land, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - MD Anderson Regional Care Center-The Woodlands, The Woodlands, Texas
  - Deke Slayton Cancer Center, Webster, Texas
  - Intermountain Medical Center, Murray, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - South Jordan Health Center, South Jordan, Utah
  - Norris Cotton Cancer Center-North, Saint Johnsbury, Vermont
  - Inova Alexandria Hospital, Alexandria, Virginia
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Augusta Health Cancer Center, Fishersville, Virginia
  - Mary Washington Hospital, Fredericksburg, Virginia
  - Sentara Cancer Institute at Sentara CarePlex Hospital, Hampton, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Roanoke, Virginia
  - Sentara Virginia Beach General Hospital, Virginia Beach, Virginia
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Overlake Hospital Medical Center, Bellevue, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Virginia Mason Federal Way Medical Center, Federal Way, Washington
  - Tacoma/Valley Radiation Oncology Centers-Gig Harbor, Gig Harbor, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Tri-Cities Cancer Center, Kennewick, Washington
  - Skagit Valley Hospital Regional Cancer Care Center, Mount Vernon, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Tacoma/Valley Radiation Oncology Centers-Puyallup, Puyallup, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Spokane Valley Cancer Center-Mayfair, Spokane, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - Tacoma/Valley Radiation Oncology Centers-Saint Joe's, Tacoma, Washington
  - Compass Oncology Vancouver, Vancouver, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Fox Valley Surgical Associates Limited, Appleton, Wisconsin
  - Radiology Associates of Appleton/ThedaCare Regional Medical Center, Appleton, Wisconsin
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Sacred Heart Hospital, Eau Claire, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Community Memorial Hospital, Menomonee Falls, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Surgical Associates of Neenah SC, Neenah, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Wheaton Franciscan Cancer Care - All Saints, Racine, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - Saint Michael's Hospital, Stevens Point, Wisconsin
  - Marshfield Clinic Stevens Point Center, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - The Alyce and Elmore Kraemer Cancer Care Center, West Bend, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
- Canada (12):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Atlantic Health Sciences Corporation-Saint John Regional Hospital, Saint John, New Brunswick
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - CIUSSSEMTL-Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - McGill University Department of Oncology, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - CHU de Quebec-L'Hotel-Dieu de Quebec (HDQ), Québec, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Ireland (2):
  - Saint Lukes Hospital, Dublin, Co Dublin
  - University College Hospital Galway, Galway, Co Galway
- Chaim Sheba Medical Center, Tel Litwinsky, Israel
- Japan (8):
  - Tohoku University School of Medicine, Sendai, Aoba-ku
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Hyogo Cancer Center, Akashi, Hyōgo
  - Iwate Medical University School of Medicine, Morioka, Iwate
  - Gunma University Hospital, Gunma, Maebashi
  - Niigata University Medical and Dental Hospital, Niigata, Niigata
  - Shikoku Cancer Center, Matsuyama
  - Saitama Medical University International Medical Center, Saitama
- San Juan City Hospital, San Juan, Puerto Rico
- Yonsei University Health System-Severance Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Mamounas EP, Bandos H, White JR, Julian TB, Khan AJ, Shaitelman SF, Torres MA, Vicini FA, Ganz PA, McCloskey SA, Lucas PC, Gupta N, Li XA, McCormick B, Smith B, Tendulkar RD, Kavadi VS, Matsumoto K, Seaward SA, Irvin WJ Jr, Lin JY, Mutter RW, Muanza TM, Stromberg J, Jagsi R, Weiss AC, Curran WJ Jr, Wolmark N. Omitting Regional Nodal Irradiation after Response to Neoadjuvant Chemotherapy. N Engl J Med. 2025 Jun 5;392(21):2113-2124. doi: 10.1056/NEJMoa2414859. PMID 40466065
- [Derived] Ferrarazzo G, Nieri A, Firpo E, Rattaro A, Mignone A, Guasone F, Manzara A, Perniciaro G, Spinaci S. The Role of Sentinel Lymph Node Biopsy in Breast Cancer Patients Who Become Clinically Node-Negative Following Neo-Adjuvant Chemotherapy: A Literature Review. Curr Oncol. 2023 Sep 25;30(10):8703-8719. doi: 10.3390/curroncol30100630. PMID 37887530
- [Derived] Ditsch N, Rubio IT, Gasparri ML, de Boniface J, Kuehn T. Breast and axillary surgery in malignant breast disease: a review focused on literature of 2018 and 2019. Curr Opin Obstet Gynecol. 2020 Feb;32(1):91-99. doi: 10.1097/GCO.0000000000000593. PMID 31833973